CLINICAL TRIAL: NCT07333534
Title: Effectiveness of Hard Tissue Augmentation With or Without Connective Tissue Graft Following Immediate Dental Implants in the Esthetic Zone: A Randomized Controlled Study
Brief Title: Hard Tissue Augmentation With or Without Connective Tissue Graft in Immediate Esthetic Implants
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Baghdad (Other)
Responsible Party: Principal Investigator, Khalid Walid Khalid, Principal Investigator, University of Baghdad
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 973124
Record Dates: First submitted 2025-12-15; First posted 2026-01-12 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2025-11

CONDITIONS: Dental Implant
Keywords: immediate implant; maxillary esthetic zone; CTG; jumping gap; bone augmentation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hard tissue augmentation with connective tissue graft (Experimental): Hard tissue augmentation (bone grafting) with additional connective tissue graft (CTG) performed at the same time following immediate dental implant in the esthetic zone
  Interventions: Procedure: Immediate dental implant in the esthetic zone
- Hard tissue augmentation (Active Comparator): Hard tissue augmentation (bone grafting) following immediate dental implant in the esthetic zone.
  Interventions: Procedure: Immediate dental implant in the esthetic zone

INTERVENTIONS:
Procedure: Immediate dental implant in the esthetic zone — Placement of immediate dental implant after tooth extraction in the maxillary esthetic zone.

SUMMARY:
This randomized controlled study is aimed to evaluate the esthetic, clinical, and radiographic outcomes following the placement of immediate single-tooth implant with hard and soft tissue augmentation.

Subjects will randomly assigned to one of two groups:

* Group A (control group) receiving an immediate single-tooth implant in the esthetic zone with bone augmentation only.
* Group B (study group) receiving an immediate single-tooth implant in the esthetic zone with bone augmentation and connective tissue graft (CTG).

The main questions it aims to answer is:

Is there is a significant difference in the esthetic outcome between bone augmentation alone and bone augmentation combined with connective tissue graft after immediate dental implant in the esthetic zone?

ELIGIBILITY:
Inclusion Criteria:

* Patients with a non-restorable tooth or a remaining root without signs of acute infection in the maxillary esthetic zone.
* The failing tooth is an incisor, canine or first bicuspid in the maxilla bounded by natural sound teeth.
* Sufficient bone (>4 mm) apically and palatally to allow for proper implant positioning with sufficient primary stability (≥35 N cm).
* Sufficient mesial-distal and interocclusal space for placement of the implant and definitive restoration.

Exclusion Criteria:

* Patients with systemic conditions affecting bone healing (e.g., uncontrolled diabetes).
* Teeth with current acute periapical infection.
* Dehiscence of the labial (facial) bone plate after extraction.
* Signs of uncontrolled periodontal disease.
* Heavy smokers and vulnerable groups (pregnant females and decision-impaired individuals).
* History of head and neck radiation therapy.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Estimated)
Dates: Start 2025-12-20 (Estimated); Primary Completion 2026-06 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
Pink Esthetic Score (PES) | Pink esthetic score (PES) will be assessed at 6 months postoperatively.
  Seven variables to be scored: mesial papilla, distal papilla, curvature of the facial mucosa, level of the facial mucosa, alveolar process, soft tissue color, and texture of facial gingiva at the implant site. A score of 0, 1, or 2 will be given to each parameter to obtain a final score of 14.

SECONDARY OUTCOMES:
Hard tissue assessment (facial bone thickness) | 6 months postoperatively
  Using Cone-Beam Computed Tomography (CBCT) to assess the thickness of the facial (labial/buccal) plate of bone at two points: the implant platform and a point 5mm apical to the implant platform.
Patient satisfaction questionnaire | 6 months postoperatively
  Assessment of patient satisfaction will be performed at 6 months postoperatively with a self-administered patient questionnaire regarding overall satisfaction and satisfaction of color and shape of the mucosa using a visual analogue scale (VAS, left = very dissatisfied [0], right = very satisfied [10].
Implant survival rate | 6 months postoperatively
  Implant survival rate at 6 months (defined by absence of mobility, infection, pain, and peri-implant bone loss).
Rate of complications | From the intervention to 6 month postoperatively
  complications such as infection, graft rejection and peri-implantitis will be assessed from the intervention up to 6 months postoperatively.

IPD SHARING:
Plan to Share IPD: Undecided